CLINICAL TRIAL: NCT00725010
Title: Temodal (TMZ) in Concomitant Radiochemotherapy Followed by Sequential TMZ Chemotherapy in Newly Diagnosed Glioblastoma Multiforme Patients - an Observational Program
Brief Title: Temozolomide in Concomitant Radiochemotherapy Followed by Sequential Temozolomide Chemotherapy - Observational Program (Study P04816)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04816
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy; Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Participants with newly diagnosed Glioblastoma multiforme who were prescribed temozolomide and radiotherapy as standard care.
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Temozolomide — Temozolomide will be administered orally at 75 mg/m^2 with radiotherapy during the concomitant treatment phase. After four weeks, temozolomide will be administered at 150 mg/m^2 to 200 mg/m^2 from Day 1 to Day 5 of six therapy cycles during the monotherapy phase.
  Other Names: Temodal; Temodar; SCH 052365
Radiation: Radiotherapy — Radiotherapy will consist of fractionated focal irradiation at a dose of 2 Gy per fraction given Monday through Friday for a total dose of 60 Gy, administered with temozolomide during the concomitant treatment phase.
  Other Names: Radiation therapy; Irradiation

SUMMARY:
The purpose of this program is to evaluate the safety, tolerability, and efficacy of the new concomitant and sequential temozolomide regimen in newly diagnosed Glioblastoma patients in a routine care setting.

DETAILED DESCRIPTION:
Participant sampling method: consecutive patient sampling.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Glioblastoma multiforme

Exclusion Criteria:

* History of hypersensitivity to temozolomide or its components, or to dacarbazine.
* Women who are pregnant or breast-feeding.
* Patients with severe myelosuppression.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with newly diagnosed Glioblastoma multiforme
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Planned Temozolomide+Radiotherapy: Subjects with newly diagnosed Glioblastoma multiforme. Temozolomide was administered orally once daily at 75 mg/m^2 with radiotherapy for 6 weeks during the concomitant treatment phase. After four weeks, temozolomide was administered at 150 mg/m^2 to 200 mg/m^2 from Day 1 to Day 5 of six therapy cycles during the monotherapy phase. Radiotherapy consisted in fractionated focal irradiation at a dose of 2 Gy per fraction given Monday through Friday for a total dose of 60 Gy, administered with temozolomide during the concomitant treatment phase.
Period: Overall Study
Arm/Group | Planned Temozolomide+Radiotherapy
Started | 50 (Only in 50 of 64 participants the documentation of therapy and follow-up was received and evaluated.)
Completed | 25
Not Completed | 25
Not completed — Toxicity | 9
Not completed — Tumor Progression | 7
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Hepatopathy probably not Temodal-related | 1
Not completed — Suspect lymph nodes neck thorax abdomen | 1
Not completed — No further documentation | 1
Not completed — Intensified treatment scheme: 3 on 1 off | 2

BASELINE CHARACTERISTICS:
Arm/Group | Planned Temozolomide+Radiotherapy
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Region of Enrollment [Number; unit: participants]
  Austria | 50

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Adverse Events in the Indicated Categories
Time Frame: Weekly during the concomitant treatment phase, and then monthly during the monotherapy phase
Measure: Number; unit: Adverse Events
Groups:
- Temozolomide+Radiotherapy: Participants with newly diagnosed Glioblastoma multiforme who received temozolomide + radiotherapy during the combined therapy phase (per-protocol treatment). Temozolomide was administered orally once daily at 75 mg/m^2 with radiotherapy for 6 weeks during the concomitant treatment phase. After four weeks, temozolomide was administered at 150 mg/m^2 to 200 mg/m^2 from Day 1 to Day 5 of six therapy cycles during the monotherapy phase. Radiotherapy consisted in fractionated focal irradiation at a dose of 2 Gy per fraction given Monday through Friday for a total dose of 60 Gy, administered with temozolomide during the concomitant treatment phase.
- Temozolomide Alone: Participants with newly diagnosed Glioblastoma multiforme treated with temozolomide alone (despite the study plan, 6 participants only received temozolomide and no radiotherapy; results are presented separately for these 6 participants). Temozolomide was administered orally once daily at 75 mg/m^2 with radiotherapy for 6 weeks. After four weeks, temozolomide was administered at 150 mg/m^2 to 200 mg/m^2 from Day 1 to Day 5 of six therapy cycles.
Arm/Group | Temozolomide+Radiotherapy | Temozolomide Alone
Number analyzed (Participants) | 44 | 6
Adverse Events
  Unlikely Related to Temozolomide | 35 | 1
  Possibly Related to Temozolomide | 14 | 0
  Probably Related to Temozolomide | 22 | 1

2. Primary Outcome: Number of Participants Who Discontinued Due to Toxicity
Time Frame: Weekly during the concomitant treatment phase, and then monthly during the monotherapy phase
Measure: Number; unit: Participants
Arm/Group | Temozolomide+Radiotherapy | Temozolomide Alone
Number analyzed (Participants) | 44 | 6
Participants | 8 | 1

ADVERSE EVENTS:
Arm/Group | Temozolomide+Radiotherapy | Temozolomide Alone
Serious Adverse Events (participants affected / at risk) | 8/44 | 1/6
Other Adverse Events (participants affected / at risk) | 12/44 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide+Radiotherapy (N=44) | Temozolomide Alone (N=6)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dural fistula (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide+Radiotherapy (N=44) | Temozolomide Alone (N=6)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No